CLINICAL TRIAL: NCT03330171
Title: Safety and Immunogenicity of Measles Vaccine, Varicella Vaccine and Hepatitis-A Vaccine in HIV-exposed and HIV-unexposed South African Children
Brief Title: Safety and Immunogenicity of Measles Vaccine, Varicella Vaccine and Hepatitis-A Vaccine
Acronym: MV/VV/Hep-AV
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Shabir Madhi, Investigator, University of Witwatersrand, South Africa
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MV/VV/Hep-AV
Record Dates: First submitted 2017-10-12; First posted 2017-11-06 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Measles; Varicella; Hepatitis A
Keywords: Immunogenicity; Safety; Vaccine
MeSH Terms: conditions — Measles; Chickenpox; Hepatitis A | interventions — Measles Vaccine; Hepatitis A Vaccines; Chickenpox Vaccine

STUDY DESIGN:
Intervention Model Description: Participants receive measles vaccine as part of routine medical care at 6 and 12 months of age. Half of the participants will receive varicella vaccine at 18 months of age and the other half will receive hepatitis-A at 18 months of age. All vaccines are administered according to their approved dosages, formulations and indications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV-unexposed children (Other): HIV-unexposed children enrolled in a randomized open label study on the pneumococcal conjugate vaccine (PCV1+1) will be invited to participate in this study. Children enrolled in the PCV1+1 study will receive all vaccines included in the South African public immunization program. Measles vaccine (0.5 mL, subcutaneous injection) will be adminstered at 6 months of age and 12 months of age. Varicella vaccine (0.5 mL, subcutaneous injection) or Hepatitis-A vaccine (0.5 mL, intra-muscular injection) will be administered to the participants at 18 months of age as an additional benefit for participating in the study.
  Interventions: Biological: Measles vaccine; Biological: Hepatitis-A vaccine; Biological: Varicella vaccine
- HIV-exposed children (Other): A cohort of HIV-exposed children will be recruited. Measles vaccine (0.5 mL, subcutaneous injection) will be adminstered at 6 months of age and 12 months of age. Varicella vaccine (0.5 mL, subcutaneous injection) or Hepatitis-A vaccine (0.5 mL, intra-muscular injection) will be administered to the participants at 18 months of age as an additional benefit for participating in the study.
  Interventions: Biological: Measles vaccine; Biological: Hepatitis-A vaccine; Biological: Varicella vaccine

INTERVENTIONS:
Biological: Measles vaccine — All participants will receive measles vaccine at 6 and 12 months of age, according to the South African immunization schedule. All study vaccines are currently licensed in South Africa and will be administered according to their approved dosages, formulations and indications.
  Other Names: Measles vaccine (MeasBio) 0.5 mL
Biological: Hepatitis-A vaccine — Half of the participants (n=135) will receive hepatitis-A vaccine at 18 months of age.
  Other Names: Hepatitis-A vaccine (Varilrix) 0.5 mL
Biological: Varicella vaccine — Half of the participants (n=135) will receive varicella vaccine at 18 months of age.
  Other Names: Varicella vaccine (Avaxim Paediatric) 0.5 mL

SUMMARY:
This trial will evaluate the safety and immunogenicity of: i) measles vaccine (CAM-70) after primary dose at 6 months (MV1) and booster vaccination at 12 months (MV2); ii) a single dose of varicella vaccination at 18 months; and iii) a single dose of hepatitis-A vaccination at 18 months in HIV-exposed and HIV-unexposed South African children.

DETAILED DESCRIPTION:
Measles vaccine (MV) can reduce childhood mortality and is currently recommended to all South African children aged 6 months. Only one study has examined the safety and immunogenicity of the recommended CAM-70 measles vaccine strain in children under 9 months of age. In addition, there are limited data on the safety and immunogenicity of varicella vaccine (VV) and Hepatitis-A vaccination (Hep-AV) in HIV-exposed and HIV-unexposed children in Sub-Saharan Africa.

This is a prospective, observational cohort study nested within a larger randomized, open-label trial on pneumococcal-conjugate vaccine (PCV) titled PCV1+1. 70 HIV-exposed and 200 HIV-unexposed children will be enrolled at Chris Hani Baragwanath Academic Hospital (CHBAH) and neighbouring primary health clinics.

Immune responses to the vaccines will be measured as rate of seroconversion, rate of seroprotection, and geometric mean titres (GMT) one month post primary immunization (MV1, VV, Hep-AV) and one month post booster dose (MV2). In addition, pre-vaccination and medium long-term antibody levels at 4.5 months, 12 months and 18 months will be evaluated. Number of adverse events in all immunized infants will be recorded throughout the study duration and compared between groups. Long-term antibody levels at 3, 4 and 5 years of age will be measured during annual follow-up visits.

This study will add to the current evidence on immunizing infants with MV (CAM-70) at 6 and 12 months of age. Data will be stratified by HIV-exposure and HIV-infection, thereby offering insight in the influence of HIV on post-vaccination immune responses. The findings on VV/Hep-AV safety, immunogenicity and seroprevalence will be useful to informing future immunization policies in Sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≤18 weeks;
2. Parent/guardian able to provide informed consent;
3. Available for the duration of the study;
4. Enrolled as a participant in the PVC1+1 trial AND born to HIV-uninfected woman; OR Born to HIV-infected mother AND infant CD4% ≥25% if HIV-infected;
5. Birth weight >2499g AND weight of >3.5 kg at time of proposed enrolment;
6. Being a healthy child (except for HIV status in HIV-exposed cohort) based on medical history and physical examination by the study staff.

Exclusion Criteria:

1. Significant major congenital abnormalities;
2. Received measles vaccination, varicella vaccination or hepatitis-A vaccination since birth;
3. Previous hospitalization for respiratory illness following discharge from hospital at birth;
4. Known allergy to vaccine components;
5. Febrile illness (axillary temperature ≥37.8°C) at time of screening;
6. Known or suspected immunodeficiency condition other than HIV;
7. Planning to relocate outside of the study area during the study period;
8. Receipt of blood transfusion or any other blood products (including immunoglobulins) since birth, receipt of such products during the course of the study will require withdrawal of the child from the study;
9. History of confirmed measles, varicella or hepatitis-A disease since birth.

Ages: 18 Weeks to 19 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 278 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with seroprotective antibody titres (IgG ≥330 mIU/ml quantified by ELISA) one month post booster measles vaccination | 13 months of age (one month post booster measles vaccine)
  Measured as seroprotection rate one month post booster measles vaccine in HIV-exposed (HEU, HIV-infected) and HIV-unexposed South African children.

SECONDARY OUTCOMES:
Number of participants with seroprotective antibody titres (IgG ≥300 mIU/ml quantified by ELISA) one month post varicella vaccination | 19 months of age (one month post vaccination)
  Measured as seroprotection rate one month post varicella immunization in HIV-exposed (HEU, HIV-infected) and HIV-unexposed South African children.
Number of participants with seroprotective antibody titres (IgG ≥20 mIU/ml quantified by ELISA) one month post hepatitis-A vaccination | 19 months of age (one month post vaccination)
  Measured as seroprotection rate one month post hepatitis-A immunization in HIV-exposed (HEU, HIV-infected) and HIV-unexposed South African children.
Number of participants with vaccine-related adverse events after primary measles vaccination | 6 months of age
  Participants will be observed for at least 30 minutes after vaccination so that clinic personnel can observe and document any potential adverse reactions to the vaccine. Report of vaccine-related local (redness, swelling, pain/tenderness, itching) and systemic (fever, vomiting, poor appetite, irritability and decreased activity) adverse events will be solicited using diary card in the 7 days after vaccination.
Number of participants with vaccine-related adverse events after booster measles vaccination | 12 months of age
  Participants will be observed for at least 30 minutes after vaccination so that clinic personnel can observe and document any potential adverse reactions to the vaccine. Report of vaccine-related local (redness, swelling, pain/tenderness, itching) and systemic (fever, vomiting, poor appetite, irritability and decreased activity) adverse events will be solicited using diary card in the 7 days after vaccination.
Number of participants with vaccine-related adverse events after varicella vaccination | 18 months of age
  Participants will be observed for at least 30 minutes after vaccination so that clinic personnel can observe and document any potential adverse reactions to the vaccine. Report of vaccine-related local (redness, swelling, pain/tenderness, itching) and systemic (fever, vomiting, poor appetite, irritability and decreased activity) adverse events will be solicited using diary card in the 7 days after vaccination.
Number of participants with vaccine-related adverse events after hepatitis-A vaccination | 18 months of age
  Participants will be observed for at least 30 minutes after vaccination so that clinic personnel can observe and document any potential adverse reactions to the vaccine. Report of vaccine-related local (redness, swelling, pain/tenderness, itching) and systemic (fever, vomiting, poor appetite, irritability and decreased activity) adverse events will be solicited using diary card in the 7 days after vaccination.
Persistence of immunogenicity | 3, 4 and 5 years of age
  Antibody concentrations and number of participants with seroprotective antibody levels to measles, varicella and hepatitis-A vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Shabir A Madhi, MD, PhD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- Chris Hani Baragwanath Academic Hospital; Nrf/Dst Vpd Rmpru, Soweto, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: No
Currently no plan to share IPD.

REFERENCES:
- [Derived] Mutsaerts EAML, van Cranenbroek B, Madhi SA, Simonetti E, Arns AJ, Jose L, Koen A, van Herwaarden AE, de Jonge MI, Verhagen LM. Impact of nutritional status on vaccine-induced immunity in children living in South Africa: Investigating the B-cell repertoire and metabolic hormones. Vaccine. 2024 May 22;42(14):3337-3345. doi: 10.1016/j.vaccine.2024.04.034. Epub 2024 Apr 17. PMID 38637212
- [Derived] Mutsaerts EAML, Nunes MC, Bhikha S, Ikulinda BT, Jose L, Koen A, Moultrie A, Grobbee DE, Klipstein-Grobusch K, Weinberg A, Madhi SA. Short-term immunogenicity and safety of hepatitis-A and varicella vaccines in HIV-exposed uninfected and HIV-unexposed South African children. Vaccine. 2020 May 8;38(22):3862-3868. doi: 10.1016/j.vaccine.2020.03.045. Epub 2020 Apr 16. PMID 32307279
- [Derived] Mutsaerts EAML, Nunes MC, Bhikha S, Ikulinda BT, Boyce W, Jose L, Koen A, Moultrie A, Cutland CL, Grobbee DE, Klipstein-Grobusch K, Madhi SA. Immunogenicity and Safety of an Early Measles Vaccination Schedule at 6 and 12 Months of Age in Human Immunodeficiency Virus (HIV)-Unexposed and HIV-Exposed, Uninfected South African Children. J Infect Dis. 2019 Sep 26;220(9):1529-1538. doi: 10.1093/infdis/jiz348. PMID 31282539